CLINICAL TRIAL: NCT02097394
Title: A Randomized Controlled Study on Combizym and Bifidobacteria to Prevent the Recurrence of Colon Polyps
Brief Title: The Clinical Study on Combizym and Bifidobacteri to Prevent the Recurrence of Colon Polyps
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, professor,chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RJYYXHNK-002
Record Dates: First submitted 2013-07-12; First posted 2014-03-27 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Combizym; Bifidobacteri; Colon Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Combizym; Pancreatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Combizym-treated group (Active Comparator): The patients who received polypectomy of colon polyps take the digestion enzyme (Combizym) regularly.
  Interventions: Drug: Combizym
- Bifidobacteri-treated group (Active Comparator): The patients who received polypectomy of colon polyps take Bifidobacteri regularly
  Interventions: Drug: Bifidobacteri
- Combizym + Bifidobacteri-treated group (Active Comparator): The patients who received polypectomy of colon polyps take drugs (Combizym + Bifidobacteri) regularly
  Interventions: Drug: Combizym + Bifidobacteri
- control (No Intervention): The patients who received polypectomy of colon polyps take no drugs

INTERVENTIONS:
Drug: Combizym — Combizym( 1 tablet, po, tid)
  Other Names: Oryz-Aspergillus Enzyme And Pancreatin Tablet; (provided by Nordmark Arzneimittel GmbH & Co. KG)
  Arms: Combizym-treated group
Drug: Bifidobacteri — Bifidobacteri (2 tablet, po, tid)
  Other Names: Live Combined Bifidobacterium，Lactobac and Enterococcus Capsules; (produced by Shanghai XinYi Company)
  Arms: Bifidobacteri-treated group
Drug: Combizym + Bifidobacteri — Combizym( 1 tablet, po, tid) + Bifidobacteri (2 tablet, po, tid)
  Other Names: Combizym(Oryz-Aspergillus Enzyme And Pancreatin Tablet); (produced by Nordmark Arzneimittel GmbH & Co. KG); Bifidobacteri(Live Combined Bifidobacterium，Lactobac and Enterococcus Capsules); (produced by Shanghai XinYi Company)
  Arms: Combizym + Bifidobacteri-treated group

SUMMARY:
The study hypothesis is whether digestion enzyme(Combizym) and intestinal flora drugs(Bifidobacteria) can decease recurrence rate of colon polyps

DETAILED DESCRIPTION:
Colon polyps has high recurrence rate in the digestion diseases. However, the reasons are not clear. The possible reasons for the recurrence of colon polyps include intestinal inflammation (e.g., Ulcerative colitis), intestinal flora imbalance (the benefit intestinal bacteria reduced, which lead to diarrhea or constipation), long-term indigestion. The investigators propose to examine whether digestion enzyme (Combizym) and intestinal flora drugs(Bifidobacteria) can decease recurrence rate of colon polyps

ELIGIBILITY:
Inclusion Criteria:

-Patients who have cutted colon polyps in one month, and the diagnosis were proved by pathological analysis

Exclusion Criteria:

* have organic or other functional disease
* pregnant or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
recurrence of colon polyps | one year
  The whole patients need be examined by colonoscopy one year later. The recurrence rate of colon polyps will be acquired in different arms

CONTACTS AND LOCATIONS:
Overall Officials: Shengliang Chen, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China